CLINICAL TRIAL: NCT04207788
Title: HIp Fracture REhabilitation Programme for Elderly With Hip Fracture
Brief Title: HIP Fracture REhabilitation Programme
Acronym: HIP-REP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carsten Bogh Juhl (Other)
Collaborators: Municipality of Herlev (Unknown); Municipality of Gentofte (Unknown); Municipality of Lyngby-Taarbaek (Unknown); Municipality of Furesoe (Unknown); Municipality of Rudersdal (Unknown); Herlev and Gentofte Hospital (Other); Jonkoping University (Other); Intersectoral Research Unit (Unknown); Metropolitan University College (Other); Danish Association of Occupational Therapist (Other); Danish Regions Development and Research (Unknown)
Responsible Party: Sponsor-Investigator, Carsten Bogh Juhl, Principal investigator, Herlev and Gentofte Hospital
Organization: Herlev and Gentofte Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-19066989
Record Dates: First submitted 2019-12-19; First posted 2019-12-23 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Hip Fractures
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Intervention Model Description: Activity-based intervention
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): HIP-REP programme offers elderly with hip fracture add on activity-focused interventions.
  Interventions: Other: HIP-REP
- Usual care (Active Comparator): The elderly with hip fracture in the control group will receive usual care.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: HIP-REP — HIP-REP programme is an add on to usual care which includes 5 add on individual activity-focused interventions that will be tailored to the need of elderly with hip fracture in a liaison with the health care professionals. Home visits and follow-up phone call will be a part of programme.
  Arms: Intervention
Other: Usual care — The elderly in the control group will receive usual rehabilitation. with a focus on mobilization within 24 hours postoperative as an in-patient. In the municipality physiotherapy is offered twice a week for approximately 12 weeks postoperative focusing on neuromotor control over hip, activation and strengthening of muscles as well as increase mobility. When relevant, the elderly receives a home visit by an occupational therapist who assess ADL behaviours, the use of assistive devices and the environmental hazards, preparing and adapting the home environment to prevent falls.
  Arms: Usual care

SUMMARY:
Objectives: To evaluate the effect of a HIP-REP on the quality and independence in ADL ability (performance), measured with the Assessment of Motor and Process Skills (AMPS) and health-related Quality of Life (QoL).

Hypothesis: The HIP-REP will increase the quality and independence in ADL performance, measured with AMPS and health-related QoL measure.

DETAILED DESCRIPTION:
Little is known about the effect of an intersectoral rehabilitation intervention aiming at reducing the decrease in Activities of Daily Living (ADL) ability for elderly with hip fractures. Despite positive surgical outcomes, one-quarter dies within a year after surgery, around eight percent are readmitted to hospital, and just one-third regain their pre-fracture level of physical functioning and ADL ability. After hip fracture, the loss of independence, and further decrease in ADL ability often persists beyond three months after surgery. This increases the risk of social isolation, depression and thus a decrease in QoL. Therefore, the investigators want to evaluate whether an activity-based rehabilitation intervention across sectors is effective and influences this fragile group of patients. The investigators hope to increase the ability to safely and independently perform ADL in elderly with hip fractures, and thereby enhance their health-related QoL.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 years or older
* Recent proximal hip fracture (S 72.0 medial femur fracture, S 72.1, pertrochanteric femur fracture, S 72.2 subtrochanteric femur fracture)
* Living at home prior to hip fracture in Herlev, Gentofte, Furesoe, Rudersdal or Lyngby-Taarbæk municipalities
* Ability to give informed consent

Exclusion Criteria:

* Not expected to be discharged to home or rehabilitation centers in the municipality
* Not able to speak and/or understand Danish
* Have prior severe physical and /or mental disabilities

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-01-28 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Assessment of Motor and Process Skills | Change frombaseline at motor and process skills 3 and 6 months after baseline testing
  The assessment measures the quality of a person's activity of daily living task performance. An observational assessment that allows for evaluation of change in motor and process skills and their effect on the ability of an individual to perform complex or instrumental and personal activities of daily living. The instrument consists of 16 motor and 20 process skill abilities that are rated on a 4-point scale. The rating scale is based on the following criteria (Quality of performance); 4 = Competent, 3 = Questionable, 2 = Ineffective or 1 = Severely deficient. In all, 36 discrete ratings of motor and process skills are made during observation.

SECONDARY OUTCOMES:
European Quality of Life Questionnaire | At baseline and 3 and 6 months after baseline testing
  A survey collecting information about health related quality of life comprising five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.
Verbal Rating Scale | At baseline and 3 and 6 months after baseline testing
  An assessment measuring the intensity of pain. The patient chooses one of those: none, mild, moderate or severe.
Functional Recovery Score | at baseline and 3 and 6 months after baseline testing
  Functional Recovery Score assess the level of function with eleven-items comprised of three main components: basic activities of daily living assessed by four items, instrumental activities of daily living assessed by six items, and mobility assessed by one item. Basic activities of daily living comprise 44 percent of the score; instrumental activities of daily living comprise 23 percent, and mobility comprises 33 percent. Complete independence in basic and instrumental activities of daily living and mobility results in a score of 100percent.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physiotherapy and Occupational Therapy, Copenhagen University Hospital, Herlev and Gentofte, Copenhagen, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fairhall NJ, Dyer SM, Mak JC, Diong J, Kwok WS, Sherrington C. Interventions for improving mobility after hip fracture surgery in adults. Cochrane Database Syst Rev. 2022 Sep 7;9(9):CD001704. doi: 10.1002/14651858.CD001704.pub5. PMID 36070134
- [Derived] Ropke A, Lund K, Thrane C, Juhl C, Morville AL. Developing an individualised cross-sectoral programme based on activities of daily living to support rehabilitation of older adults with hip fracture: a qualitative study. BMJ Open. 2021 Jun 18;11(6):e044539. doi: 10.1136/bmjopen-2020-044539. PMID 34145009

DOCUMENTS (1):
  • Statistical Analysis Plan (2021-04-21): https://cdn.clinicaltrials.gov/large-docs/88/NCT04207788/SAP_000.pdf